CLINICAL TRIAL: NCT06949800
Title: Probiotics to Treat HSIL and Reduce Persistent High Risk HPV Infection in Women and Men Living With HIV
Brief Title: CASCADE 2002: PROTECT Study, "PRObiotics to TrEat Anal preCancer Trial
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Exegi Pharma, LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25361; U54CA242646 (NIH)
Record Dates: First submitted 2025-04-22; First posted 2025-04-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: HSIL, High Grade Squamous Intraepithelial Lesion; HPV-Related Squamous Cell Carcinoma; Anal HSIL
Keywords: HIV; Anal intraepithelial neoplasia (AIN) 3; p16+ AIN 2
MeSH Terms: conditions — Squamous Intraepithelial Lesions | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Blinded: EXE-346 probiotic (Experimental): Participants will be blinded and stratified on gender and according to hrHPV status (HPV16 present or absent in baseline swab). After confirmation of biopsy-proven HSIL, participants will receive sachets of EXE-346 or placebo, with the contents suspended in water and consumed orally twice per day for 3 months (12 weeks) with follow-up visits at 24 and 36 weeks. Participants will undergo High resolution anoscopy (HRA) as a safety check at Visit 3 (12 weeks) and at Visit 4 (24 weeks) to ensure HRA has not progressed to cancer. Biopsies will only be performed if there is any concern for progression. Participants with active HSIL at week 36 will be treated with non-investigational, standard of care, hyfrecation as soon as possible, but within 8 weeks.
  Interventions: Drug: EXE-346 Probiotic; Procedure: Usual Care High Resolution Anoscopy (HRA)
- Blinded: Placebo (Placebo Comparator): Participants will be blinded and stratified on gender and according to hrHPV status (HPV16 present or absent in baseline swab). After confirmation of biopsy-proven HSIL, participants will receive sachets of EXE-346 or placebo, with the contents suspended in water and consumed orally twice per day for 3 months (12 weeks) with follow-up visits at 24 and 36 weeks. Participants will undergo High resolution anoscopy (HRA) as a safety check at Visit 3 (12 weeks) and at Visit 4 (24 weeks) to ensure HRA has not progressed to cancer. Biopsies will only be performed if there is any concern for progression. Participants with active HSIL at week 36 will be treated with non-investigational, standard of care, hyfrecation as soon as possible, but within 8 weeks.
  Interventions: Drug: Placebo; Procedure: Usual Care High Resolution Anoscopy (HRA)

INTERVENTIONS:
Drug: EXE-346 Probiotic — Given as a single-dose, powder packet to mix with water
  Other Names: EXE-346 Probiotic formula; Probiotic
  Arms: Blinded: EXE-346 probiotic
Drug: Placebo — Given as a single-dose, powder packet to mix with water
  Other Names: Blinded Placebo
  Arms: Blinded: Placebo
Procedure: Usual Care High Resolution Anoscopy (HRA) — Non-investigational HRA will be performed
  Other Names: HRA

SUMMARY:
This study is focused on treatment of anal high-grade squamous intraepithelial lesions (HSIL) in persons with HIV (PWH), with the ultimate goal of applying the approach toward prevention of anal cancer in this population

DETAILED DESCRIPTION:
This is a randomized double-blinded, placebo-controlled trial.

PRIMARY OBJECTIVES:

I. Evaluate regression to no disease among people with HIV (PWH) with anal HSIL at baseline at Week 36.

II. To determine the safety of EXE-346 in PWH.

SECONDARY OBJECTIVES:

I. To evaluate regression to LSIL or normal at Week 36 among PWH with anal HSIL at baseline.

II. To evaluate clearance at Week 36 to HPV-negative in anal swab for type(s) found at the baseline visit in PWH.

EXPLORATORY OBJECTIVES:

I. To determine if changes in the microbiome from baseline to Week 36 correlate with regression of anal HSIL to low grade squamous intraepithelial lesions (LSIL) or normal, or clearance of HPV found at baseline.

Participants will be randomized in a block design used to stratify women or men according to high-risk human papillomavirus (hrHPV) status (HPV16 present or absent in baseline swab). After confirmation of biopsy-proven HSIL, participants will receive sachets of EXE-346 or placebo for up to 3 months (12 weeks) with follow-up visits at 24 weeks and 36 weeks. Participants with HSIL at week 36 may be treated with non-investigational, standard of care, hyfrecation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Participant in ULACNet-101 or participant screened specifically for ULACNet-102.
3. Biopsy-proven anal HSIL (men or women) shown as part of participation in the ULACNet-101 study or at a screening visit for ULACNet-102.
4. At least one focus of anal HSIL must be large enough to be monitored for response, i.e.,not completely removed after the screening biopsy.
5. Total volume of HSIL is less than 50% of the anal canal or perianal region.
6. Must be actively on treatment with effective antiretroviral therapy (ART) regimen for at least three months preceding enrollment (Visit 1, Day 1) in ULACNet-101 or at screening for ULACNet-102.
7. HIV RNA <200 copies/ml at baseline.
8. Cluster of differentiation 4 (CD4) nadir above 200 cells per microliter (uL)
9. Eastern Cooperative Oncology Group (ECOG) performance status <=1 (Karnofsky >= 70%).
10. Participants must meet the following laboratory parameters within 3 months before enrollment:

    1. Leukocytes: ≥3,000/mm^3.
    2. Absolute neutrophil count: ≥1,500/mm^3.
    3. Platelets: ≥100,000/mm^3.
    4. Elevation of aspartate aminotransferase (AST), alanine aminotransferase (ALT), or bilirubin <2 times the upper limit of normal.
11. Not pregnant or breast feeding and one of the following:

    1. Of non-childbearing potential (i.e. persons aged 60 years or older or who have had a hysterectomy or tubal ligation or are postmenopausal, as defined by no menses for at least 12 months and without an alternative medical cause).
    2. Persons aged less than 60 years of childbearing potential and agree to practice highly effective contraception from initiation of taking EXE-346 or placebo through 14 days after taking the last dose of EXE-346 or placebo. Highly effective methods of contraception include one or more of the following:

    i.Male partner who is sterile (medically effective vasectomy) prior to the female participant's entry into the study and is the sole sexual partner for the female participant.

ii.Hormonal (oral, intravaginal, transdermal, implantable or injectable); Progestogen-only hormonal contraceptives without inhibition of ovulation are not considered to be highly effective.

iii. An intrauterine hormone-releasing system. iv. An intrauterine device. v. Bilateral tubal occlusion or removal. vi. Sexual abstinence, only if the participant refrains from heterosexual intercourse from initiation taking EXE-346 or placebo through 14 days after taking the last dose of EXE-346 or placebo and it is the usual lifestyle of the participant.

Exclusion Criteria:

1. History of any anogenital cancer.
2. Presence of untreated cervical HSIL or cervical cancer.
3. Anal HSIL on clinical examination or biopsy that clinicians are concerned for cancer.
4. Receipt of chemotherapy, radiotherapy or immunosuppressive medication in three months preceding enrollment in ULACNet-101 or at the screening visit for ULACNet-102.
5. Immunosuppression as a result of underlying illness or treatment including:

   1. Use of high dose corticosteroids (>10 mg/day prednisone or equivalent) for >=7 days (inhaled, otic, topical and ophthalmic corticosteroids are permitted).
   2. Primary immune deficiency disease.
   3. Use of synthetic or biologic disease-modifying anti-rheumatic drugs.
   4. History of bone marrow or solid organ transplant.
   5. History of any other clinically significant autoimmune or immunosuppressive disease.
6. Participant initiated a new treatment with antibiotics within the 2 weeks prior to screening or plans to start antibiotic therapy during the study period.
7. Participant is taking NSAIDs as a long-term treatment (ie, consistent use for at least 4 days/week each month). Acute use of NSAIDs is allowed.
8. Participant has known hypersensitivity to EXE-346 or any product components.
9. Current known infection with severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
10. Warts so extensive that they preclude the clinician from determining the extent and location of HSIL.
11. Sustained, manually confirmed, sitting systolic blood pressure >150 mm Hg or <90 mm Hg or a diastolic blood pressure >95 mm Hg as measured by 3 readings taken 15 minutes apart at screening or Visit 1.
12. History of significant thrombocytopenia, history of thrombosis with thrombocytopenia (TTS) syndrome or heparin-induced thrombocytopenia.
13. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
14. Participant has participated in any clinical study of an approved or unapproved investigational medicinal product within the 30 days prior to screening.
15. Any other finding that, in the opinion of the Investigator deems the participant unsuitable for the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with no disease present | Up to 36 weeks
  No anal disease defined as complete regression of lesions as determined by examination of biopsies obtained at HRA
Proportion of participants reporting treatment-emergent adverse events | Up to 36 weeks
  The frequency of participants reporting adverse events by group will be classified according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0

SECONDARY OUTCOMES:
Proportion of participants with demonstrated disease regression | Up to 36 weeks
  Regression of HSIL associated with any hrHPV type to LSIL or lower, as determined by examination of biopsies obtained at HRA
Proportion of participants with HPV-negative status | 1 day
  The proportion of participants with HPV-negative on anal swab for type(s) found at baseline will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Palefsky, MD, Principal Investigator — University of California, San Francisco
Locations (2):
- University of California, San Francisco, San Francisco, California, United States
- University of Puerto Rico Comprehensive Cancer Center, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
De-identified information will be shared with study collaborators
Supporting Information: Study Protocol, SAP, ICF
Time Frame: For the duration of study activities